CLINICAL TRIAL: NCT00496522
Title: Phase II Evaluation of Proton Beam Therapy for Skull Base Chondrosarcoma
Brief Title: Proton Beam Therapy for Chondrosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0915; NCI-2012-01510 (Registry Identifier: NCI CTRP-Clinical Trials Reporting Registry)
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chondrosarcoma
Keywords: Skull Base Chondrosarcoma; Proton Beam Therapy; Chondrosarcoma; CNS
MeSH Terms: conditions — Chondrosarcoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Proton Beam Therapy (Other): Proton Beam Therapy - A total dose of up to 70 CGE given at 2.0 CGE per daily fraction for 35 fractions.
  Interventions: Procedure: Proton Beam Therapy

INTERVENTIONS:
Procedure: Proton Beam Therapy — A total dose of up to 70 CGE given at 2.0 CGE per daily fraction for 35 fractions.

SUMMARY:
The goal of this clinical research study is to learn if proton beam therapy, with or without photon beam radiation therapy, is effective in the treatment of skull base chondrosarcoma. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Patients who have skull base chondrosarcoma require complicated treatment because of its challenging location and nearness to critical structures within the brain.

Pathology will be confirmed prior to discussion of the study.

If you are found to be eligible to take part in this study, you will receive proton beam therapy, no sooner than 2 weeks after the last surgery to remove tumor. You will receive proton beam therapy once a day for about 35 treatments (7 weeks). Treatment will be given for 5 days in a row each week (except for Saturdays, Sundays, and holidays) at the Proton Center in Houston. The whole process should take up to 1 hour each day.

If your doctor feels it is necessary, the proton beam therapy may be combined with standard photon therapy.

After the proton beam, and possibly photon beam, therapy, you will be asked to come in for study follow-up visits every year, until the study is completed. At these visits, you will have magnetic resonance imaging (MRI) scans, blood draws (less than 1 teaspoon) to monitor your pituitary function, and neuropsychological testing. For the neuropsychological testing, you will be interviewed and tested by a neuropsychologist to evaluate your memory, fluency (the ability to talk and form words) complex thinking ability, planning ability, and coordination. These tests could last from 1-2 hours. You will also have eye exams performed by an ophthalmologist from MD Anderson and hearing exams. It is anticipated that it will take about 5 years to complete this study.

This is an investigational study. The proton beam center and its treatment are approved by the FDA for patient use. A total of up to 15 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed Grade 1-3 chondrosarcoma of the skull base
2. Contrast enhanced postop MRI or CT if there is clinical contraindication for MRI of the skull base obtained with 90 days of study registration at M. D. Anderson
3. The patient has been assessed by MDACC skull base surgeons to have undergone maximal surgical debulking of disease
4. Karnofsky Performance status greater than or equal to 60
5. Signed informed consent

Exclusion Criteria:

1. Previous irradiation of the skull base
2. Documented evidence of disseminated metastatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04-28 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Time to Local Recurrence | Baseline to local recurrence (evaluation every six months during estimated 5 year study)
  Local recurrence defined as progression on magnetic resonance imaging (MRI) or CT if MRI is contraindicated.

CONTACTS AND LOCATIONS:
Overall Officials: David Grosshans, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org